CLINICAL TRIAL: NCT05359770
Title: Effects of an Inspiratory Muscle Training Protocol Associated With Neurological Stimulation by HD-tDCS on the Diaphragmatic Cortex in Post-COVID-19 Subjects
Brief Title: Association of Inspiratory Muscle Training With HD-tDCS for Assistance to Patients With Long Covid-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Suellen Marinho Andrade (Other)
Responsible Party: Sponsor-Investigator, Suellen Marinho Andrade, Principal Investigator, Federal University of Paraíba
Organization: Federal University of Paraíba (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FUniversity of Paraíba
Record Dates: First submitted 2022-03-22; First posted 2022-05-04 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Coronavirus; Inspiratory Muscle Training; Respiratory Infection; COVID-19
Keywords: Transcranial direct current stimulation; Non-invasive brain stimulation; Inspiratory muscle training; Functional capacity; Maximal inspiratory pressure
MeSH Terms: conditions — Coronavirus Infections; Respiratory Tract Infections; COVID-19 | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Experimental: Experimental Group/ Active HD-tDCS Patients randomly enrolled in this group will receive 10 sessions of anodal HD-tDCS stimulation on cortical representation zone of left diaphragmatic motor cortex associated to respiratory training; for 20 minutes (each session) with a 2mA intensity. The electrical current will be delivered with a ramp-up time of 30 s, held at 3mA for 20 min, and then ramped down over 30 s.
  Interventions: Device: Active HD-tDCS; Device: Control group
- Sham Comparator (Sham Comparator): Sham Comparator: Control Group / Sham Group In the sham condition, the device will provide a 30-second ramp-up followed immediately by a 30-second ramp down in HD-tDCS associated with inspiratory muscle training for 20 minutes
  Interventions: Device: Active HD-tDCS; Device: Control group

INTERVENTIONS:
Device: Active HD-tDCS — Experimental group: 10-sessions of anodal HD-tDCS ( tDCS 1x1, developed by Soterix Medical Inc.) associated to respiratory training; for 20 minutes (each session). It will be delivered a 3mA intensity electrical current accordingly 10/20 International System on cortical representation zone of left diaphragmatic motor cortex using HD-tDCS.
Device: Control group — Sham Control: 10-sessions of anodal HD-tDCS( tDCS 1x1, developed by Soterix Medical Inc.) associated to respiratory training; for 20 minutes (each session) with a 3mA intensity. The device will provide a 30-second ramp-up followed immediately by a 30-second ramp down.
  Other Names: Sham control

SUMMARY:
COVID-19 is an infectious disease which presents a heterogenous clinical presentation. Recent investigations suggest that people who were infected by COVID-19 often develop physical disabilities (i.e. pain, fatigue), neurological complications and and mainly disorders of the respiratory system, such as respiratory muscle weakness after hospital discharge. Many therapeutic approaches such as transcranial direct current stimulation (tDCS) have been proposed to minimize functional and structural impairments. The aim of the present study is to evaluate the effects of inspiratory muscle training associated with stimulation of the diaphragmatic motor cortex through hd-tdcs in post-COVID-19 patients on inspiratory muscle strength, pulmonary function, inflammatory levels and functional capacity.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had a medical diagnosis of COVID-19, clinically stable, able to respond to simple commands, able to walk for six minutes and who sign study consent form will be enrolled.

Exclusion Criteria:

* Those who present associated neurological diseases, pregnant, users of psychoactive drugs, patients who have metallic implants, electronic devices, pacemakers, or epileptic patients will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-09-22 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
Maximal inspiratory pressure | From date of randomization (2 weeks before intervention beginning) and up to 10 weeks (T1)
  Maximal inspiratory pressure response to inspiratory muscle training in association with diaphragmatic motor cortex neurostimulation

SECONDARY OUTCOMES:
Functional capacity | From date of randomization (2 weeks before intervention beginning) and up to 10 weeks (T1)
  Compare baseline to treatment responses in the distance covered on the 6-minute walk test (6MWT). Its measurement has focused on the examination on a broader health indicator than morbidity, as it is correlated with quality of life.
Forced vital capacity (FVC), forced expiratory volume 1st second (FEV1) and peak expiratory flow (PEF) by spirometry | From date of randomization (2 weeks before intervention beginning) and up to 10 weeks (T1)
  Data of pulmonary function given by FCV, FEV1 and PEF will be assessed before and after pulmonary responses using spirometry
Inflammatory biomarkers | From date of randomization (2 weeks before intervention beginning) and up to 10 weeks (T1)
  Correlate levels of inflammatory markers (interleukin-6 and C-reactive protein) with inspiratory muscle training and/or diaphragmatic motor cortex neurostimulation
Body composition by bioelectrical impedance | From date of randomization (2 weeks before intervention beginning) and up to 10 weeks (T1)
  Body composition analysis (body fat composition, muscle mass composition, body mass index) will be carried out by bioelectrical impedance analysis
Depression level with Hamilton Anxiety Rating Scale (score 0 to 58) | From date of randomization (2 weeks before intervention beginning) and up to 10 weeks (T1)
  Anxiety level will be evaluate through Hamilton Anxiety Rating Scale which measures the severity of anxiety symptoms in a score 0 to 58. In current practice, it is accepted that scores greater than 25 points characterize severely depressed patients, scores between 18 and 24 points characterize moderately depressed patients, and scores between 7 and 17 points characterize patients with mild depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Suellen Andrade, pHD, João Pessoa, Paraíba, Brazil